CLINICAL TRIAL: NCT04400175
Title: Effects on Coordination of Sucking, Swallowing and Breathing Process of a Valved Feeding System in Late-preterm Newborns. The Safe Oral Feeding Trial (SOFT)
Brief Title: Effects of a Valved Feeding System in Late-preterm Newborns: the Safe Oral Feeding Trial
Acronym: SOFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Cresi, MD, PhD, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOFT-study
Record Dates: First submitted 2020-04-25; First posted 2020-05-22 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Premature Birth; Feeding; Difficult, Newborn; Feeding, Bottle
Keywords: late-preterm newborns, valved feeding system
MeSH Terms: conditions — Premature Birth; Bottle Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-ESP (Experimental): B-ESP group will be fed with a feeding system with a valved ergonomic teat.
  Interventions: Device: Valved ergonomic teat
- B-STD (Sham Comparator): B-STD will be fed with a standard feeding system.
  Interventions: Device: Standard silicon teat

INTERVENTIONS:
Device: Valved ergonomic teat — Administration of milk with a feeding system with a valved ergonomic teat in late preterm newborns.
  Arms: B-ESP
Device: Standard silicon teat — Administration of milk with a feeding system with a standard silicon teat
  Arms: B-STD

SUMMARY:
Comparing with a randomized controlled trial two different feeding systems in two groups of late-preterm newborns for evaluating which is more efficient in promoting the coordination in the process of sucking-swallowing-breathing and better cardiorespiratory stability.

The B-ESP group will be fed with a feeding system with a valved ergonomic teat; the B-STD with a standard feeding system.

DETAILED DESCRIPTION:
The swallowing patterns are still immature in the newborn, especially if preterm. An incomplete synchronization in the process of sucking, swallowing and breathing could lead to some difficulty during feedings with desaturations and risk of milk inhalation in the upper airway tract. Moreover, a dysfunctional or immature pattern of sucking, swallowing and breathing also affect the post-prandial period, tiring the newborn and increasing the cardio-respiratory instability.

Breastfeeding promote the development of a physiological coordination of the process of sucking, swallowing and breathing, guaranteeing high and stable values of oxygenation during feedings. On the other hand, bottle-feeding could be responsible of a difficult coordination among the phases of swallowing and breathing. In an healthy, at term, brestfed newborn is observed a typical pattern of sucking-swallowing-expiration with a ratio of 1:1:1. In a bottlefed newborn this ratio is 2-12:1:4, with a relative increase of the period of sucking compared to the swallowing one, that could lead to apnoeas and desaturations.

The differences between the two feedings modality are more accentuated in the late-preterm newborn, which is more prone to cardio-respiratory instability compared to the healthy at term newborn, because of the immaturity of the respiratory centers in the brainstem, and of the processes responsible for the coordination of the sucking, swallowing and breathing .

However breastfeeding, in spite of the fact that is crucial for the development of the correct process of sucking, can be challenging in the premature infant because it requires a considerable physical effort.

Therefore, disposing of devices for nutrition able to facilitate oral feeding, simulating the physiologic breastfeeding, is necessary. In this way, we can contribute to the development of the proper sucking-swallowing-breathing pattern and to improve cardio-respiratory stability.

In literature there are multiple studies carried out on term newborns demonstrating the importance of the negative pressure or air vacuum created in the oral cavity, in order to promote the emptying of the lactiferous ducts and/or of the teat and simultaneously promote the maintainance of the right respiratory pattern. An ergonomic feeding system with a valve able to create vacuum could be able to respond to the demands of late preterm newborns.

Aim of the study is to evaluate the effects of a trial with an experimental feeding system with a teat with a valve able to facilitate the vacuum in the oral cavity on the pattern of sucking-swallowing and breathing in late preterm newborns.

NUMBER OF PATIENTS Precise data regarding swallowing/respiration rate in bottle-fed late preterm infants in the first 3 days of life are lacking in the literature. Considering a mean swallow/respiration ratio of 1.5 and a variance of 0.5, obtained from surveys performed at our center prior to the study, a sample size of 38 infants per arm was estimated to achieve 80% power to detect a 30% difference on the primary outcome with a significance level of 0.05.

STUDY DESIGN Late preterm newborns eligible to enter in the study, prior obtaining the informed consent from parents, will be assigned in the "B-ESP" or "B-STD" group through a process of block randomisation, controlled by a software.

Newborns included in the randomisation, after a training of 3 meals with the feeding bottle assigned from the randomisation, can be entered in the study.

Newborns included in the study will be monitored for the entire duration of a meal and the subsequent 3-hours period. This monitoring will be collected in two different times (T1 and T2): in the second day of life (24-48 hours of life) and in the fourth day of life (72-96 hours of life). The study includes an audio recording of the swallowings through a microphone in the room and the recordings of the process of sucking and swallowing through a cutaneous sensor.

In addition, a cardiorespiratory monitoring with a poligraph will be made, considering oxygen saturation, cardiac and respiratory frequency and electrocardiography. The meal's video recording will permit a subsequent classification of the sucking movements and the evaluation of any possible interference in the polygraphic recording.

FEEDING DEVICES

Newborns of the B-STD group will be fed using a classic disposable feeding device, which is actually in use in our centre and provided by our hospital, composed of:

* a 150 mL feeding bottle in polypropylene, devoid of BPA;
* a silicon teat, devoid of BPA, available in two types, (a slow graduated flow and a standard flow) depending on the necessities and suction abilities of the baby;
* a protective plug.

Newborns of the B-ESP group will be fed using a feeding system with a valved ergonomic teat, composed of:

* a slow-flow ergonomic silicon teat
* polipropilene bottle with a capacity of 150 mL, with a ventilation valve on the bottom
* silicon valve

Newborns will be fed with defined quantities of maternal milk or bank donated milk, based on weight and gestational age.

The meal will be administered by the caregiver (a parent or a nurse) previously trained. The meal's administration will be performed keeping the baby in the caregivers's arms in the ESL position (semielevated side-lying). At the end of the feeding process the newborn will be repositioned in his cradle in the supine position.

The cardiosaturimetric evaluation will be performed using a system of polygraphic monitoring, which allows a simultaneous non-invasive recording of cardiorespiratory parameters, noises and movements associated to the sucking and swallowing processes combined to video recordings.

The evaluation of the sucking process will be carried out using a structured questionnaire composed by 31 items, which allows to distinguish normal suction (mature) from disorganized and dysfunctional ones.

Considering simultaneously the cardiosaturimetric parameters, video, audio and cutaneous sensor's recordings, it is possible to obtain a more accurate evaluation of the processes of swallowing, sucking and breathing of the newborn during meal administration. It is also possible to identify the exact moment of the breathing process assigned to the newborn's swallowing.

CLINICAL DATA

At birth:

* gestational age;
* weight in grams;
* z-score;
* sex;
* type of delivery;
* peri-partum condition, including possible administration of prenatal corticosteroids;
* type of support provided at birth;

At T1 and T2:

* hours from birth;
* weight;
* z-score;
* number of meals in a day;
* type of milk administered;
* overall volume administered expressed in mL in a day;
* duration of a meal expressed in minutes;
* number of regurgitation or vomit during the administration of a meal;
* number of regurgitation or vomit after the admninistration of a meal;

At discharge:

* weight;
* z-score;
* number of meals in a day;
* type of feeding (exclusive breastfeeding; exckusive bottlefeeding or mixed)
* overall volume administered expressed in mL in a day;

INSTRUMENTAL DATA

* Number of suctions;
* Number of swallowings;
* Number of apnoeas;
* Average duration of apnoeas;
* Number of oxygen desaturations
* Minimal oxygen saturation;
* Number of reduction of cardiac frequency (bradycardia);
* Minimal cardiac frequency. The definition of apnoea, oxygen desaturation and bradycardia applied in this study are the ones defined by literature (Di Fiore JM, Arko MK, Miller MJ, et al. Cardiorespiratory Events in Preterm Infants Referred for Apnea Monitoring Studies. PEDIATRICS. 2001;108(6):1304-1308.)
* APNOEA: arrest of the breathing acts for a period of at least 20 seconds or arrest of the breathing acts for a period of at least 5 seconds associated with bradycardia and/or desaturations;
* OXYGEN DESATURATIONS: reduction of the oxygen saturation (SpO2) <80% or of at least 5% compared to the baseline, for at least 4 seconds.
* BRADYCARDIA: reduction of the cardiac frequency under 80 bpm for at least 4 seconds

STATISTICAL ANALYSIS

Statistical analysis will be carried out using the STATISTICA software package for Windows (StatSoft, Inc., Tulsa, Oklahoma, USA). Every newborn in the experimental group will be matched with a newborn of the control group similar for gestational age and weight. For the normal distribution, data will be tested with the Kolmogorov-Smirnov test and with the exploratory data analysis. Data will be expressed as statistical mean and standard deviation (SD) or as median and interquantile range depending on the relative distribution. The differences between the polisonnographic data will be evaluated with the Student's T test or through a similar non-parametric test depending on the distribution: Fisher test for comparison between categorical data and regression tests (linear and non-linear) for comparison between continuous variables. Statistical significance is set as p<0.05.

EXPECTED RESULTS

The more physiological administration of milk with a feeding system with a valved ergonomic teat, could better promote the development of coordination in the process of sucking-swallowing-breathing. Therefore inhalation and cardiosaturimetric events during a meal and immediately after will be reduced and therefore the newborn's oral feeding tolerance will increase, making it more similar to physiological breastfeeding.

Bottle-feeding milk administration with a feeding system with a valved ergonomic teat in the first days of life, the period when exclusive breastfeeding is more difficult, could also promote the transition between bottle-feeding to breastfeeding, because this mechanism is more similar to the physiological one.

If the results of this study will support this hypotesis, feeding system with a valved ergonomic teat could be chosen as a non-pharmacological treatment for late-preterm newborns who encounter difficulty in the oral feeding, such as cardio-respiratory instability during the sucking process and risk of milk inhalation when the breastfeeding is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 34+0 - 36+6 weeks at birth;
* Exclusive oral feeding;
* Bottle-feeding for at least a meal a day;

Exclusion Criteria:

* Newborns with exclusive breastfeeding;
* Newborns with congenital anomalies, perinatal asphyxia, respiratory or neurological issues, genetic syndromes, infections, metabolic diseases;
* Ongoing administration of medication able to interfere with esophageal or respiratory function;
* Newborns who require respiratory support, including oxygen-therapy via nasal-cannula;
* Newborns who require oral or nasal feeding tube;

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluating the level of coordination in the sucking-swallowing-breathing pattern in the B-ESP group compared with the B-STD | Calculated throughout 72 hours
  This evaluation will be recorded at 24 and 72 hours of life and defined from the suckings/swallowings ratio.
  The literature describes this parameter as strongly associated to a higher maturity of the sucking-swallowing-breathing pattern; in fact, a ratio of sucking-swallowing-breathing of 1:1:1 describes the mature pattern, typical of the breastfeeding and considered the optimum for a newborn.

SECONDARY OUTCOMES:
Coefficient of variation of time between sucking and swallowing | Calculated throughout 72 hours
  This coefficient is expressed in seconds. a lower coefficient corresponds to breastfeeding
Mean percentage of incidence of breaths that precede and follow the swallowings | Calculated throughout 72 hours
  This percentage is classified by Lau et al. (the average interval between two breathing acts monitored during a meal of an healthy at term newborn varies between 1.2-2 seconds)
Evaluation of the sucking processes | Calculated throughout 72 hours
  This evaluation is made through the a structured questionnaire composed by 31 items
Evaluation of cardiorespiratory stability | Calculated throughout 72 hours
  This evaluation is made considering frequency and characteristics of cardiorespiratory events (during and after meal administration)
Evaluation of meal tolerance | Calculated throughout 72 hours
  This evaluation is carried out considering the number of vomiting and regurgitations during and after the meal, volume in mL per meal, number of meals per day
Number of breastfed newborns at the time of dimission | Calculated throughout 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cresi, MD; PhD, Principal Investigator — Città della Salute e della Scienza - Ospedale S.Anna - University of Turin
Locations (1):
- Città della Salute e della Scienza - Ospedale S.Anna - University of Turin, Turin, Italy

REFERENCES:
- [Background] Joshi R, van Pul C, Sanders A, Weda H, Bikker JW, Feijs L, Andriessen P. A Strategy to Reduce Critical Cardiorespiratory Alarms due to Intermittent Enteral Feeding of Preterm Neonates in Intensive Care. Interact J Med Res. 2017 Oct 20;6(2):e20. doi: 10.2196/ijmr.7756. PMID 29054835
- [Background] Poets CF, Langner MU, Bohnhorst B. Effects of bottle feeding and two different methods of gavage feeding on oxygenation and breathing patterns in preterm infants. Acta Paediatr. 1997 Apr;86(4):419-23. doi: 10.1111/j.1651-2227.1997.tb09034.x. PMID 9174231
- [Background] Gross RD, Trapani-Hanasewych M. Breathing and Swallowing: The Next Frontier. Semin Speech Lang. 2017 Apr;38(2):87-95. doi: 10.1055/s-0037-1599106. Epub 2017 Mar 21. PMID 28324898
- [Background] Chen CH, Wang TM, Chang HM, Chi CS. The effect of breast- and bottle-feeding on oxygen saturation and body temperature in preterm infants. J Hum Lact. 2000 Feb;16(1):21-7. doi: 10.1177/089033440001600105. PMID 11138220
- [Background] Goldfield EC, Richardson MJ, Lee KG, Margetts S. Coordination of sucking, swallowing, and breathing and oxygen saturation during early infant breast-feeding and bottle-feeding. Pediatr Res. 2006 Oct;60(4):450-5. doi: 10.1203/01.pdr.0000238378.24238.9d. Epub 2006 Aug 28. PMID 16940236
- [Background] Simmer K, Kok C, Nancarrow K, Hepworth AR, Geddes DT. Novel feeding system to promote establishment of breastfeeds after preterm birth: a randomized controlled trial. J Perinatol. 2016 Mar;36(3):210-5. doi: 10.1038/jp.2015.184. Epub 2015 Dec 10. PMID 26658121
- [Background] Mizuno K, Ueda A. Changes in sucking performance from nonnutritive sucking to nutritive sucking during breast- and bottle-feeding. Pediatr Res. 2006 May;59(5):728-31. doi: 10.1203/01.pdr.0000214993.82214.1c. PMID 16627890
- [Background] Mathew OP. Respiratory control during nipple feeding in preterm infants. Pediatr Pulmonol. 1988;5(4):220-4. doi: 10.1002/ppul.1950050408. PMID 3237449
- [Background] Ward, N. Feeding and Swallowing Disorders in Infancy: Assessment and Management. J. Hum. Lact. 11, 147-147 (1995)
- [Background] Sakalidis VS, Geddes DT. Suck-Swallow-Breathe Dynamics in Breastfed Infants. J Hum Lact. 2016 May;32(2):201-11; quiz 393-5. doi: 10.1177/0890334415601093. Epub 2015 Aug 28. PMID 26319112
- [Background] Dalgleish SR, Kostecky LL, Blachly N. Eating in "SINC": Safe Individualized Nipple-Feeding Competence, a Quality Improvement Project to Explore Infant-Driven Oral Feeding for Very Premature Infants Requiring Noninvasive Respiratory Support. Neonatal Netw. 2016;35(4):217-27. doi: 10.1891/0730-0832.35.4.217. PMID 27461200
- [Background] Whyte R. Safe discharge of the late preterm infant. Paediatr Child Health. 2010 Dec;15(10):655-66. doi: 10.1093/pch/15.10.655. PMID 22131865
- [Background] Meier P, Patel AL, Wright K, Engstrom JL. Management of breastfeeding during and after the maternity hospitalization for late preterm infants. Clin Perinatol. 2013 Dec;40(4):689-705. doi: 10.1016/j.clp.2013.07.014. Epub 2013 Sep 21. PMID 24182956
- [Background] Lau C. Development of infant oral feeding skills: what do we know? Am J Clin Nutr. 2016 Feb;103(2):616S-21S. doi: 10.3945/ajcn.115.109603. Epub 2016 Jan 20. PMID 26791183
- [Background] Geddes DT, Sakalidis VS, Hepworth AR, McClellan HL, Kent JC, Lai CT, Hartmann PE. Tongue movement and intra-oral vacuum of term infants during breastfeeding and feeding from an experimental teat that released milk under vacuum only. Early Hum Dev. 2012 Jun;88(6):443-9. doi: 10.1016/j.earlhumdev.2011.10.012. Epub 2011 Nov 26. PMID 22119233
- [Background] Cannon AM, Sakalidis VS, Lai CT, Perrella SL, Geddes DT. Vacuum characteristics of the sucking cycle and relationships with milk removal from the breast in term infants. Early Hum Dev. 2016 May;96:1-6. doi: 10.1016/j.earlhumdev.2016.02.003. Epub 2016 Mar 8. PMID 26964010
- [Background] da Costa SP, van der Schans CP, Zweens MJ, Boelema SR, van der Meij E, Boerman MA, Bos AF. The development of sucking patterns in preterm, small-for-gestational age infants. J Pediatr. 2010 Oct;157(4):603-9, 609.e1-3. doi: 10.1016/j.jpeds.2010.04.037. Epub 2010 Jun 14. PMID 20542296
- [Background] Fucile S, McFarland DH, Gisel EG, Lau C. Oral and nonoral sensorimotor interventions facilitate suck-swallow-respiration functions and their coordination in preterm infants. Early Hum Dev. 2012 Jun;88(6):345-50. doi: 10.1016/j.earlhumdev.2011.09.007. Epub 2011 Sep 29. PMID 21962771
- [Background] Lau C, Smith EO, Schanler RJ. Coordination of suck-swallow and swallow respiration in preterm infants. Acta Paediatr. 2003 Jun;92(6):721-7. PMID 12856985